CLINICAL TRIAL: NCT00709280
Title: Infant Study of Inhaled Saline in Cystic Fibrosis
Acronym: ISIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CF Therapeutics Development Network Coordinating Center (Network)
Collaborators: Cystic Fibrosis Foundation (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ISIS002; U01HL092931 (NIH); U01HL092932 (NIH)
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; hypertonic saline; inhaled saline
MeSH Terms: conditions — Cystic Fibrosis | interventions — Saline Solution, Hypertonic; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active treatment group (Experimental): 7% Hypertonic Saline administered via inhalation twice daily for 48 ± 4 weeks
  Interventions: Drug: 7% Hypertonic Saline (HS)
- Control group (Active Comparator): 0.9% Isotonic Saline administered via inhalation twice daily for 48 ± 4 weeks
  Interventions: Drug: 0.9% Isotonic Saline (IS)

INTERVENTIONS:
Drug: 7% Hypertonic Saline (HS) — Administered via inhalation twice daily for 48 ± 4 weeks. The delivery system is a PARI Sprint Junior nebulizer with a PARI Baby face mask or mouthpiece driven by a PARI Pro Neb compressor.
  Other Names: Hyper-Sal™, inhaled saline
  Arms: Active treatment group
Drug: 0.9% Isotonic Saline (IS) — Administered via inhalation twice daily for 48 ± 4 weeks. The delivery system is a PARI Sprint Junior nebulizer with a PARI Baby face mask or mouthpiece driven by a PARI Pro Neb compressor.
  Other Names: Normal saline
  Arms: Control group

SUMMARY:
The purpose of this study is to assess whether 7% hypertonic saline (HS) is an effective and safe therapy in infants and young children with CF.

DETAILED DESCRIPTION:
A growing body of evidence supports the importance of intervention in Cystic Fibrosis (CF) lung disease during infancy and early childhood, in order to potentially delay or prevent irreversible lung disease. Yet, aside from antimicrobial therapies, the CF community has no clinical trial evidence base with which to guide pulmonary therapies in children <6 years of age. Hypertonic Saline (HS) is the most attractive chronic maintenance therapy to investigate in these young children because it addresses defective mucociliary clearance, an early step in the cascade of events leading to CF lung disease that is expected to be abnormal prior to the onset of airway infection and inflammation.

This study is a randomized, parallel group, controlled trial to assess the efficacy and safety of 7% HS inhaled twice daily for 48 weeks among young children with CF 4 to < 60 months of age at enrollment. The primary hypothesis is that, compared to isotonic saline (IS), HS will decrease the number of protocol-defined pulmonary exacerbations during the 48 week treatment period. The results of the proposed trial may for the first time provide evidence for early initiation of HS, which, by improving mucociliary clearance, may delay or hinder the cycle of infection and inflammation responsible for progressive airway damage in CF lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF by newborn screening or at least one clinical feature of CF, AND either: (a) A documented sweat chloride ≥ 60 mEq/L by quantitative pilocarpine iontophoresis or (b) A genotype with two identifiable CF-causing mutations
* Informed consent by parent or legal guardian
* Age 4 months to < 60 months at Enrollment visit. If participating in Infant Pulmonary Function testing (selected sites), age 4 months to < 16 months at Enrollment visit.
* Ability to comply with medication use, study visits, and study procedures as judged by the site investigator

Exclusion Criteria:

* Acute intercurrent respiratory infection, defined as an increase in cough, wheezing, or respiratory rate with onset in 1 week preceding Enrollment visit
* Acute wheezing at Enrollment visit (prior to HS test dose), or at Infant PFT visit (prior to infant pulmonary function testing), as applicable
* Oxygen saturation < 95% (< 90% in centers located above 4000 feet elevation) at Enrollment visit (prior to HS test dose) or at Infant PFT visit (prior to infant pulmonary function testing), as applicable
* Other major organ dysfunction, excluding pancreatic dysfunction
* Physical findings that would compromise the safety of the subject or the quality of the study data as determined by the site investigator
* Investigational drug use within 30 days prior to Enrollment visit, or within 30 days prior to Infant PFT visit as applicable
* Treatment with inhaled hypertonic saline at any concentration within 30 days of Enrollment visit, or within 30 days prior to Infant PFT visit as applicable
* Chronic lung disease not related to CF
* Intolerance of test dose of HS at Enrollment visit
* A sibling that has been randomized and is still enrolled in ISIS002

Additional Exclusion Criteria for Participation in Infant Pulmonary Function Testing:

* History of adverse reaction to sedation
* Clinically significant upper airway obstruction as determined by the Site Investigator (e.g. severe laryngomalacia, markedly enlarged tonsils, significant snoring, diagnosed obstructive sleep apnea)
* Severe gastroesophageal reflux, defined as persistent frequent emesis despite anti-reflux therapy
* Acute intercurrent respiratory infection, defined as an increase in cough, wheezing, or respiratory rate with onset in 2 weeks preceding visit

Ages: 4 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 321 (Actual)
Dates: Start 2009-04; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The rate of protocol-defined pulmonary exacerbations requiring treatment with oral, inhaled or intravenous antibiotics between subjects randomized to HS and IS | during the 48 week treatment period

SECONDARY OUTCOMES:
Symptoms by parent home questionnaire administered weekly | during the 48 week treatment period
Health-related quality of life as assessed by scores from Cystic Fibrosis Questionnaire-Revised Parent Report (CFQ-R), administered quarterly | over the 48 week treatment period
Standardized cough score assessed at study visits | during the 48 week treatment period
Change in weight, height, resting respiratory rate, and room air oxygen saturation | over the 48 week treatment period
Among participants from whom Pseudomonas aeruginosa (Pa) and other CF pathogens were not isolated from respiratory cultures prior to enrollment, the proportion from whom these organisms are isolated from clinically collected respiratory cultures | measured at baseline and at 48 weeks
Pulmonary function indices measured at baseline and 48 weeks in infants 4 to 15 months of age at enrollment participating in infant pulmonary function testing (N = 100, selected sites) | over the 48 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Davis, MD, Principal Investigator — University of North Carolina, Chapel Hill; Margaret Rosenfeld, MD, MPH, Principal Investigator — Children's Hospital and Regional Medical Center; Felix Ratjen, MD, PhD, Principal Investigator — University of Toronto Hospital for Sick Children
Locations (30):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Stanford University / Lucile S. Packard Children's Hospital, Palo Alto, California
  - The Children's Hospital, Aurora, Colorado
  - Children's Memorial Hospital and Northwestern University, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Johns Hopkins University / Johns Hopkins Hospital, Baltimore, Maryland
  - University of Michigan / C.S. Mott Children's Hospital, Ann Arbor, Michigan
  - Children's Hospitals and Clinics of Minnesota, Minneapolis, Minnesota
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - University of Nebraska, Omaha, Nebraska
  - Women and Children's Hospital of Buffalo, Buffalo, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Pulmonary Division, Columbus, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia - Pediatric Respiratory Medicine, Charlottesville, Virginia
  - Children's Hospital & Regional Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - BC Children's Hospital, Vancouver, British Columbia
  - Hospital For Sick Children, Toronto, Ontario

REFERENCES:
- [Result] Rosenfeld M, Ratjen F, Brumback L, Daniel S, Rowbotham R, McNamara S, Johnson R, Kronmal R, Davis SD; ISIS Study Group. Inhaled hypertonic saline in infants and children younger than 6 years with cystic fibrosis: the ISIS randomized controlled trial. JAMA. 2012 Jun 6;307(21):2269-77. doi: 10.1001/jama.2012.5214. PMID 22610452
- [Derived] Subbarao P, Stanojevic S, Brown M, Jensen R, Rosenfeld M, Davis S, Brumback L, Gustafsson P, Ratjen F. Lung clearance index as an outcome measure for clinical trials in young children with cystic fibrosis. A pilot study using inhaled hypertonic saline. Am J Respir Crit Care Med. 2013 Aug 15;188(4):456-60. doi: 10.1164/rccm.201302-0219OC. PMID 23742699